CLINICAL TRIAL: NCT03725241
Title: Does Daily Supplementation With Glutathione Alter Immunity, Upper Respiratory Tract Infection, and Oxidative Stress in Individuals Training for a Half Marathon Race
Brief Title: Effects of Glutathione on Immunity in Individuals Training for a Marathon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas, Denton, TX (Other)
Collaborators: Kirin Holdings Company, Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18-100
Record Dates: First submitted 2018-10-05; First posted 2018-10-31 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Healthy
MeSH Terms: interventions — Glutathione

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Intervention: Dietary Supplement: Placebo supplement
  Interventions: Dietary Supplement: Placebo Supplement
- Experimental: Glutathione (Experimental): Intervention: Dietary Supplement: Glutathione supplement
  Interventions: Dietary Supplement: Glutathione Supplement

INTERVENTIONS:
Dietary Supplement: Glutathione Supplement — 1000 mg/day Glutathione
  Other Names: L-Glutathione reduced
  Arms: Experimental: Glutathione
Dietary Supplement: Placebo Supplement — Crystalline cellulose
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to determine the effects of glutathione supplement on the immune cell response and symptomatology of upper respiratory health, and antioxidant capacity in healthy people in exercise-induced model.

DETAILED DESCRIPTION:
A minimum of 60 individuals will be recruited and enrolled to complete the entire protocol in a randomized, double-blinded, 18 week placebo-controlled trial. Subjects will receive either a placebo or glutathione while participating in a stepwise exercise approach that mixes periods of high and low training volume to train subjects and improve running efficiency. Upper Respiratory Tract Infection-related health conditions will be monitored and assessed throughout the study period. Blood and saliva samples will be collected at baseline, and before and after timed 15k and half marathon runs at 12 and 16 weeks respectively.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, male or female.
* Between the ages of 19-45 years.
* Have no medical restrictions and no health conditions that would inhibit participant from marathon run.
* Be willing and able to comfortably abstain from any food supplements.
* Not participating as a subject in another study.

Exclusion Criteria:

* BMI < 20.0 or > 28.5.
* Current or prior use of tobacco products or other inhaled substance.
* More than a moderate intake of alcohol (>1 drink per day in women; >2 drinks per day in men).
* Metabolic or inflammatory disease.
* Excellent fitness based on the American College of Sports Medicine criteria for VO2max based on age and gender.
* Recent weight loss of >10 pounds in the last 3-months.
* Daily intake of ibuprofen, acetaminophen, aspirin, polyphenol supplements, multivitamins, and/or antioxidant supplements.
* Actively attempting (or planning) to lose or gain weight and/or alter body composition.
* Currently taking cholesterol-lowering medications.
* Currently taking prescription anti-inflammatory medications.
* Currently using mouthwash on a regular basis (>4 times per week).
* Orthopedic problems that would limit running capacity.
* Currently in very poor or poor fitness.
* Highly aerobic exercise trained.
* Pregnant or planning to become pregnant during the study period.
* Breast feeding
* Currently taking blood pressure medications.
* Contraindications to strenuous exercise.
* Anemic (blood hemoglobin <10 g/dL and/or hematocrit <35%).
* Diagnosed with asthma or other lung disease.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Complete Blood Count (CBC) | Evaluated at baseline, week 12 and week 16
  CBC will be drawn and white blood cell count will be evaluated as an indicator of infection.
Change in Erythrocyte Sedimentation Rate (ESR) | Evaluated at baseline, week 12 and week 16
  ESR will be measured as a marker of systematic inflammation
Change in mucosal immunity | Evaluated at baseline, week 12 and week 16
  Salivary Immunoglobulin concentrations will be tracked as a marker of the bodies ability to mount a first line defense against viruses and other pathogens
Change in T-cell population | Evaluated at baseline, week 12 and week 16
  Shifts in the T-cell concentration and population phenotypes will be tracked as a marker for readiness to fight infection
Change in T-cell response to Group A Streptococci Antigen | Evaluated at baseline, week 12 and week 16
  Measurements will provide insight regarding the in vitro capacity of the body to respond to the most common virus causing URTI

SECONDARY OUTCOMES:
Survey based tracking of upper respiratory tract infection symptoms | Continuous for 18 weeks
  Tracking of symptoms allows for calculation of % healthy vs % sick days
Incident specific tracking of upper respiratory tract infections (URTI) | Continuous for 18 weeks
  Incidence tracking of URTI allows for evaluation of comparative number, severity and recovery time from URTI
Changes in Thiobarbituric acid reactive substances (TBARs) | Evaluated at baseline, week 12 and week 16
  TBARs are a direct index of the state of lipid peroxidation which is a marker of oxidative stress
Changes in Glutathione (GSH)/Glutathione disulfide (GSSG) ratio in blood | Evaluated at baseline, week 12 and week 16
  The ratio of reduced glutathione to oxidized glutathione will be analyzed as a marker of oxidative stress and antioxidant capacity

CONTACTS AND LOCATIONS:
Overall Officials: Brian K McFarlin, PhD, Principal Investigator — University of North Texas, Denton, TX
Locations (1):
- University of North Texas, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: No